CLINICAL TRIAL: NCT06670950
Title: A Two-Part Study Investigating the Relative Bioavailability and the Potential Food Effect After a Single Oral Dose Administration of a New Formulation of SYT-510, and the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Multiple Oral Dose Administration of SYT-510 in Healthy Subjects
Brief Title: A Phase 1 Single Dose and Multiple Ascending Dose Study to Assess the Relative Bioavailability, Food Effect, Safety, Tolerability and Pharmacokinetics of SYT-510 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Synendos Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYN510CT02; 1010456 (Registry Identifier: IRAS ID)
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Relative bioavailability and food effect (Experimental): Randomised, open label, single-dose, three period, three-sequence crossover study to evaluate the relative bioavailability (rBA) of a new oral formulation of SYT-510 under fasting conditions and the effect of food in healthy participants.
  Interventions: Drug: SYT-510
- Part 2: Multiple Ascending Dose (Experimental): Randomised, double-blind, placebo-controlled multiple ascending dose (MAD) study in healthy participants to assess the safety, tolerability and pharmacokinetics (PK) of SYT-510 after repeated administrations.
  Interventions: Drug: SYT-510; Drug: Placebo

INTERVENTIONS:
Drug: SYT-510 — Oral formulation A fasted
Drug: SYT-510 — Oral formulation B fasted
  Arms: Part 1: Relative bioavailability and food effect
Drug: SYT-510 — Oral formulation A fed
  Arms: Part 1: Relative bioavailability and food effect
Drug: Placebo — Oral formulation
  Arms: Part 2: Multiple Ascending Dose

SUMMARY:
Part 1 aims to investigate the relative bioavailability of a new formulation and to assess potential food effects following oral administration of SYT-510. Part 1 will then guide dosing in Part 2, a multiple dose study which aims to assess safety, tolerability and pharmacokinetic of multiple SYT-510 administrations.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential (WOCBP) aged 18 to 65 years old (inclusive) at the date of signing the informed consent form (ICF).
* Normal ECG, showing no clinically relevant deviations, as judged by the investigator.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, at Screening and Admission (e.g Day -1 or Day -2) and a minimum weight of 50kg.

Exclusion Criteria:

* Current or recurrent disease that as judged by the Investigator may interfere with the execution of the conduct of the study.
* Laboratory parameters outside of the laboratory normal range.
* Positive test results for alcohol or drugs of abuse.
* Treatment with an investigational drug within 90 days preceding the first dose of trial medication.
* Known or suspected intolerance or hypersensitivity to the investigational product, any closely related compound, or any of the stated ingredients.
* History of significant allergic reactions (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
* Current smokers and those who have smoked within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female participants of non-childbearing potential
Enrollment: 90 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Concentration (Cmax) of SYT-510 | Up to 72 hours post-dose
Part 1: Area under the concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC0-tlast) of SYT-510 | Up to 72 hours post-dose
Part 1: AUC of SYT-510 | Up to several days post last dose
Part 2: Incidence and severity of treatment related adverse event, including abnormal laboratory events to evaluate the safety and tolerability profile of multiple ascending doses of SYT-510 | Up to Day 20

SECONDARY OUTCOMES:
Part 1: Incidence and severity of treatment related adverse event, including abnormal laboratory events to evaluate the safety and tolerability profile of single doses of SYT-510 | Up to Day 4
Part 2: Maximum observed concentration (Cmax) of SYT-510 | Up to Day 14
Part 2: Time of maximal plasma concentration (tmax) of SYT-510 | Up to Day 14
Part 2: AUCtau of SYT-510 | Up to Day 14
Part 2: Terminal elimination half-life (t1/2) of SYT-510 | Up to several days post last dose
Part 2: Accumulation ratio of SYT-510 | Up to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No